CLINICAL TRIAL: NCT01985724
Title: A Multicenter Randomized Study Comparing the Dose Dense, G-CSF-supported Sequential Administration of FE75C Followed by Docetaxel Versus Docetaxel/Cyclophosphamide Doublet as Adjuvant Chemotherapy in Women With HER-2 Negative, Axillary Lymph Node Positive Breast Cancer
Brief Title: Sequential Administration of FE75C and Docetaxel Versus Docetaxel/Cyclophosphamide in HER-2 Negative, Node Positive Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/07.17
Record Dates: First submitted 2013-11-09; First posted 2013-11-15 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Breast Cancer
Keywords: Early breast cancer; Axillary node positive; HER-2 negative; Adjuvant chemotherapy; Dose dense; Docetaxel; FEC
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Epirubicin; Cyclophosphamide; Fluorouracil; Granulocyte Colony-Stimulating Factor; Lenograstim; pegfilgrastim

ARMS (2):
- A (Active Comparator): FEC -> TXT
  Interventions: Drug: Docetaxel; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: 5-fluoruracil; Drug: Granulocyte-colony stimulating growth factor
- B (Experimental): Docetaxel/Cyclophosphamide (TC)
  Interventions: Drug: Docetaxel; Drug: Cyclophosphamide; Drug: Granulocyte-colony stimulating growth factor

INTERVENTIONS:
Drug: Docetaxel — ARM A: Docetaxel 75 mg/m2 as an IV infusion over 1h on day 1 every 2 weeks for 4 cycles ARM B: Docetaxel 75 mg/m2 as an IV infusion over 1h on day 1 every 3 weeks for 6 cycles
  Other Names: Taxotere
Drug: Epirubicin — ARM A: Epirubicin 75 mg/m2 IV push on day 1 every 2 weeks for 4 cycles
  Other Names: Farmorubicin
  Arms: A
Drug: Cyclophosphamide — ARM A: Cyclophosphamide 500 mg/m2 IV push on day 1 every 2 weeks for 4 cycles ARM B: Cyclophosphamide 600 mg/m2 IV push on day 1 every 3 weeks for 6 cycles
  Other Names: Endoxan
Drug: 5-fluoruracil — ARM A: 5-fluoruracil 500 mg/m2 IV push on day 1 every 2 weeks for 4 cycles
  Other Names: 5-FU
  Arms: A
Drug: Granulocyte-colony stimulating growth factor — rhG-CSF 5 μg/kg/d on days 3-10 after each cycle
  Other Names: Granocyte; Neulasta

SUMMARY:
In this trial investigators propose to assess the dose dense, G-CSF supported sequential administration of 4 cycles of FEC followed by 4 cycles of docetaxel versus 6 cycles of docetaxel/cyclophosphamide as adjuvant chemotherapy in women with HER-2 negative, axillary lymph node positive breast cancer

DETAILED DESCRIPTION:
Anthracycline-containing regimens are recommended as adjuvant treatment for women with node positive breast cancer. At least five large randomized clinical trials demonstrated that the addition or sequential administration of a taxane (paclitaxel or docetaxel) to an anthracycline-based regimen resulted in superior clinical outcome for women with node positive or high risk node-negative early breast cancer. In two large randomized studies the dose dense administration with G-CSF support of anthracycline-based and paclitaxel combination was superior to the same regimen administered every three weeks without growth factors as adjuvant therapy in women with axillary node positive breast cancer. In one randomized trial, docetaxel was proved superior to paclitaxel in women with metastatic breast cancer.

Data from at least one trial suggest that four cycles of a non-anthracycline but taxane-containing adjuvant regimen (docetaxel plus cyclophosphamide) provide outcomes that are at least as good, if not better than four cycles of doxorubicin/cyclophosphamide combination.

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically-confirmed unilateral invasive ductal or lobular breast adenocarcinoma
* Within 60 days after the surgical excision of the primary tumor with tumor-free operation margins; at least 10 axillary lymph nodes have to be removed.
* Tumor involvement of at least one axillary lymph node
* Absence of any clinical or radiological evidence of local or metastatic disease
* Premenopausal or postmenopausal women aged 18-75 years old
* Adequate bone marrow function (absolute neutrophil count >1500/mm3, platelet count >100.000/mm3, hemoglobin >10gr/mm3)
* Adequate liver (bilirubin <1.0 times upper limit of normal and SGOT/SGPT <2.5 times upper limit of normal) and renal function (creatinine <1.5mg/dl)
* Adequate cardiac function (LVEF>50%)
* Written informed consent

Exclusion Criteria:

* Positive pregnancy test.
* Psychiatric illness or social situation that would preclude study compliance.
* Other concurrent uncontrolled illness.
* Prior or concurrent antineoplastic therapy e.g. hormonal therapy, radiation therapy, chemotherapy, biological agents.
* Previous history of other invasive malignancy other than non-melanomatous skin cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2007-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
3-year disease-free survival | 3 years

SECONDARY OUTCOMES:
Overall survival | 3 years
Recurrence rate | Relapses by the time of 3-years follow up

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Mavrudis, MD, Principal Investigator — University Hospital of Crete
Locations (10):
- Greece (10):
  - University Hospital of Crete, Heraklion, Crete
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - "IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - "Marika Iliadis" Hospital of Athens, Dep of Medical Oncology, Athens
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - State General Hospital of Larissa, Dep of Medical Oncology, Larissa
  - "Metaxa's" Anticancer Hospital of Piraeus, 1st Dep of Medical Oncology, Piraeus
  - "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki

REFERENCES:
- [Derived] Mavroudis D, Matikas A, Malamos N, Papakotoulas P, Kakolyris S, Boukovinas I, Athanasiadis A, Kentepozidis N, Ziras N, Katsaounis P, Saloustros E, Georgoulias V; Breast Cancer Investigators of the Hellenic Oncology Research Group (HORG), Athens, Greece. Dose-dense FEC followed by docetaxel versus docetaxel plus cyclophosphamide as adjuvant chemotherapy in women with HER2-negative, axillary lymph node-positive early breast cancer: a multicenter randomized study by the Hellenic Oncology Research Group (HORG). Ann Oncol. 2016 Oct;27(10):1873-8. doi: 10.1093/annonc/mdw274. Epub 2016 Aug 8. PMID 27502729